CLINICAL TRIAL: NCT06697639
Title: Study on the Effect of WAFF Pelvic and Abdominal Mechanics Exercises During the Puerperium on Postpartum Pelvic Floor Rehabilitation for Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1-24PJ1196
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Floor Dysfunctions
Keywords: postpartum woman; puerperium; pelvic floor muscle repair

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rehabilitation Group (Experimental): In addition to routine postpartum care, small-sized WAFF air cushions will be issued during the hospitalization period to guide patients in performing the WAFF pelvic-abdominal mechanical rehabilitation exercises. Patients will also be instructed to join the experimental group's WeChat group. After discharge, researchers will upload WAFF pelvic-abdominal mechanical rehabilitation instructional videos. Patients are required to complete their rehabilitation exercises twice daily, each session lasting 10-15 minutes. Patients need to upload their exercise videos twice a week, and researchers will provide motion guidance based on the video content until the patient's postpartum follow-up examination. The abdominal rectus muscle, pelvic floor muscle function, and adherence to rehabilitation exercises will be assessed for patients in both groups at 6-8 weeks and 6 months postpartum.
  Interventions: Behavioral: Rehabilitation Group
- Control Group (No Intervention): During hospitalization, routine postpartum education and discharge instructions will be provided, including the distribution of promotional brochures and guidance on performing puerperium recovery exercises. Patients will be instructed to join the control group's WeChat group. After discharge, researchers will upload instructional videos for the recovery exercises and urge patients to perform the postpartum recovery exercises twice daily, each session lasting 10-15 minutes. Patients are required to upload their exercise videos twice a week, and researchers will provide motion guidance based on the video content until the patient's postpartum follow-up examination.

INTERVENTIONS:
Behavioral: Rehabilitation Group — In addition to routine postpartum care, small-sized WAFF air cushions will be issued during the hospitalization period to guide patients in performing the WAFF pelvic-abdominal mechanical rehabilitation exercises. Patients will also be instructed to join the experimental group's WeChat group. After discharge, researchers will upload WAFF pelvic-abdominal mechanical rehabilitation instructional videos. Patients are required to complete their rehabilitation exercises twice daily, each session lasting 10-15 minutes. Patients need to upload their exercise videos twice a week, and researchers will provide motion guidance based on the video content until the patient's postpartum follow-up examination. The abdominal rectus muscle, pelvic floor muscle function, and adherence to rehabilitation exercises will be assessed for patients in both groups at 6-8 weeks and 6 months postpartum.
  Arms: Rehabilitation Group

SUMMARY:
Ethics Review Committee, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences

Currently, in order to improve women's health throughout their entire life cycle, postpartum rehabilitation for parturients has received significant attention.

Currently, clinical postpartum rehabilitation mostly adopts a combined treatment of Kegel exercises, physical electrical stimulation, and biofeedback therapy. Kegel exercises can be applied during the puerperium. However, studies have found that some parturients find it difficult to locate the muscle contraction sensation during exercise, resulting in poor technique and effectiveness; furthermore, the training process is boring and difficult to maintain. Physical electrical stimulation and biofeedback therapy have significant therapeutic effects, but this treatment should be initiated after the puerperium and requires hospital visits, often leading to discontinuation due to long distances and time-consuming commutes.

Many experts domestically and internationally have stated that earlier postpartum rehabilitation leads to better outcomes. However, studies show that only a small percentage of patients are aware of the correct timing for postpartum rehabilitation and are able to undergo rehabilitation exercises during the puerperium. Most current studies initiate postpartum rehabilitation training from 6 to 8 weeks postpartum, with relatively few reports on pelvic and abdominal muscle training during the puerperium.

Therefore, we have introduced French WAFF pelvic and abdominal mechanical exercises and applied them to the rehabilitation of women during the puerperium. WAFF pelvic and abdominal mechanical exercises are safer, more precise, and more convenient, utilizing the instability created by the WAFF air cushion to stimulate patients' self-regulatory movements, thereby achieving a tighter core and deeper muscle groups to improve training efficiency.

Currently, the application of WAFF pelvic and abdominal mechanical exercises in China is still in the preliminary exploratory stage, and a unified and mature rehabilitation model has not yet been established. This study aims to explore the effectiveness of applying WAFF pelvic and abdominal mechanical exercises during the puerperium to improve postpartum rectus abdominis diastasis and pelvic floor dysfunction. It provides a basis for establishing a new model of puerperium rehabilitation and improving continuous obstetrical nursing.

ELIGIBILITY:
Inclusion Criteria:

* primipara
* Singleton pregnancy
* With full cognitive and behavioral abilities, and voluntarily participating

Exclusion Criteria:

* Neonate with a birth weight of >4000g
* Second-degree or higher perineal tear
* Poor healing of perineal wounds
* Individuals with severe hypertension, impaired cardiopulmonary function, and neurological diseases
* History of previous pelvic floor disorders and urogenital surgeries
* Individuals engaging in other exercises such as yoga during the puerperium

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
"Pelvic floor muscle rehabilitation status" | Prepartum；Postpartum 6-8 weeks
  PFDI-20 Pelvic Floor Distress Inventory score: It consists of a total of 20 questions related to recent bladder, bowel, and pelvic symptoms. Participants are asked to select the degree of impact these symptoms have on their lives. Each selection is scored on a scale of 0 to 4, with a total possible score ranging from 0 to 80. A higher score indicates a greater impact on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No